CLINICAL TRIAL: NCT03879941
Title: Repair of Thumb Defect by Using the Toe Nail Flap: Biomechanical Analysis of Donor Foot ,a Retrospective Cohort Study
Brief Title: Repair of Thumb Defect by Using the Toe Nail Flap
Acronym: RTDUTNF
Status: Completed | Type: Observational
Sponsor: Hebei Medical University (Other)
Collaborators: Tangshan Worker's Hospital (Other); The Second Hospital of Tangshan (Other)
Responsible Party: Principal Investigator, Chunjie Liu, Principal Investigator, Hebei Medical University
Other Study IDs: 2013-01-3
Record Dates: First submitted 2019-03-13; First posted 2019-03-19 (Actual); Last update posted 2019-03-19 (Actual); Status verified 2019-03

CONDITIONS: Thumb Injury
Keywords: Amputation; thumb reconstruction; toe transfer; foot morbidity; biomechanics

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The thumb accounts for 50% of the total hand function. This study reports the functional outcomes and complications of people with traumatic thumb amputations who underwent toe-to-thumb reconstruction.From 2013-01 to 2018-01, 29 patients with second-degree thumb defect underwent thumb reconstruction with distal phalangeal braided toenail flap. The footscan foot pressure gait analysis system was used to measure the index changes of the same foot before and after one, three and six months. The contact area, peak pressure, impulse value, contact time of each gait phase, centre of gravity coordinate and foot balance were analysed statistically. Twenty-nine cases of thumb reconstruction recovered well. After following up for 6-15 months, the appearance of the reconstructed thumb was close to normal, and the sensation was restored to S3+. The two-point discrimination was 6-8 mm, and the function of the thumb was good. The function of the donor foot was well restored, and no skin ulceration, pain and claudication were noted during walking. Compared with that before operation, the biomechanical indices of the donor foot were basically restored to normal six months after operation. Only the stress and impulse values of the third metatarsal head were significantly increased, forming a stress concentration area centred on the third metatarsal head.This study confirmed that the toe nail flap with distal phalangeal bone restored the second-degree thumb defect without destroying the main functional structure of the sole. The biomechanical indices of the donor foot were basically restored to normal six months after operation. Only the stress concentration area centred on the third metatarsal head, and the pain on the forefoot was induced after the operation. Discomfort, callus formation, metatarsal fasciitis, etc. can lead to fatigue fracture of the third metatarsal bone in severe cases, which requires further follow-up and observation.

ELIGIBILITY:
Inclusion Criteria:

1. patients with second-degree thumb defect；
2. without any foot disease or deformity before injury；
3. Written informed consent to undergo the surgical procedure；

Exclusion Criteria:

1. Concomitant phalanx fractures or other injuries needing immobilization；
2. Loss of skin substance requiring grafts or flaps
3. Uncompensated diabetes, neoplasia, haemocoagulative alterations, psychic disorders
4. Smokers

Ages: 17 Years to 46 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: The causes of injury were as follows: 2 cases of amputation and loss, 21 cases of machine rolling damage, 5 cases of rotational tear and replantation failure and 1 case of childhood traumatic defect. The patients included 19 males and 10 females with age of 17-46 years (mean 29.1 years), height of 156-179 cm (average 170.4 cm), weight of 50-80 kg (average 62.3 kg) and foot length of 23-26 cm (average 24.5 cm). The defect cases included 12 on the left side of the toe and 17 on the right side.
Sampling Method: Non-Probability Sample
Enrollment: 29 (Actual)
Dates: Start 2013-03-01 (Actual); Primary Completion 2018-03-01 (Actual); Study Completion 2018-06-01 (Actual)

PRIMARY OUTCOMES:
The contact area | Six months
  According to the anatomical region, the plantar was divided into eight stress regions.The increase or decrease of contact area reflects the stress distribution of sole after operation.
Peak pressure | Six months
  Its increase indicates that the pressure in the unit area increases when the sole touches the ground.
Impulse value | Six months
  Impulse value refers to the product of touchdown time and pressure in each stress area of the foot in each cycle. The increase of impulse is more suggestive of fatigue damage and subsequent foot deformities.
Contact time of each gait phase | Six months
  The increase or decrease it reflects the stress distribution of sole after operation.
Foot balance | Six months
  Foot balance refers to the difference of compressive stress between the inside and the outside of the foot at a certain time.

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Foucher G. Second toe-to-finger transfer in hand mutilations. Clin Orthop Relat Res. 1995 May;(314):8-12. PMID 7634655
- [Background] Pet MA, Ko JH, Vedder NB. Reconstruction of the traumatized thumb. Plast Reconstr Surg. 2014 Dec;134(6):1235-1245. doi: 10.1097/PRS.0000000000000716. PMID 25255109
- [Background] Sabapathy SR, Venkatramani H, Bhardwaj P. Reconstruction of the thumb amputation at the carpometacarpal joint level by groin flap and second toe transfer. Injury. 2013 Mar;44(3):370-5. doi: 10.1016/j.injury.2013.01.012. Epub 2013 Jan 20. PMID 23340236
- [Background] Lee KS, Chae IJ, Hahn SB. Thumb reconstruction with a free neurovascular wrap-around flap from the big toe: long-term follow-up of thirty cases. Microsurgery. 1995;16(10):692-7. doi: 10.1002/micr.1920161007. PMID 8676733
- [Background] Woo SH, Yoo MJ, Paeng JW. Recent Advances in Immediate Toe-to-Hand Transfer. J Hand Surg Asian Pac Vol. 2016 Oct;21(3):292-9. doi: 10.1142/S2424835516400099. PMID 27595944
- [Background] Buldt AK, Allan JJ, Landorf KB, Menz HB. The relationship between foot posture and plantar pressure during walking in adults: A systematic review. Gait Posture. 2018 May;62:56-67. doi: 10.1016/j.gaitpost.2018.02.026. Epub 2018 Feb 23. PMID 29524798
- [Derived] Liu C, Liu L, Liu G, Tian S, Bai J, Yu K, Tian D. Repair of thumb defect by using the toenail flap: biomechanical analysis of donor foot-a retrospective cohort study. J Orthop Surg Res. 2019 Sep 2;14(1):287. doi: 10.1186/s13018-019-1330-7. PMID 31477182